CLINICAL TRIAL: NCT02888002
Title: Internet-based vs Face-to-face Treatment for Alcohol Dependence: A Randomised, Controlled Non-inferiority Trial
Brief Title: Internet-based vs Face-to-face Treatment for Alcohol Dependence
Acronym: IMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Anne H Berman, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014/1758-31/2-2
Record Dates: First submitted 2016-01-17; First posted 2016-09-02 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Alcohol Abuse; Alcohol Dependence; Harmful Alcohol Use; Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Ethanol; Motivational Interviewing; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet-based treatment (Experimental): "Guide to better alcohol habits online". An Internet-based treatment program with online counselor support.
  Interventions: Behavioral: Guide to better alcohol habits
- Face-to-face treatment (Experimental): "Guide to better alcohol habits F2F": Face-to-face treatment with 5 individual counselor sessions at the clinic.
  Interventions: Behavioral: Guide to better alcohol habits

INTERVENTIONS:
Behavioral: Guide to better alcohol habits — A 5-module therapeutic program wich includes self-help material in printed or web-based form with interactive exercises. The program includes instructions for the therapist.
  Other Names: Motivational Interviewing (MI); Cognitive Behavioral Therapy (CBT); Behavioral Self-Control Training; eChange

SUMMARY:
A brief treatment program (MI/CBT) via face-to-face or via internet is tested in association with an outpatient addictions clinic.

DETAILED DESCRIPTION:
A 5-module program based on motivational interviewing (MI) and cognitive behavioral therapy (CBT) is tested among help-seekers at one outpatient clinic within the Stockholm Center for Dependency Disorders: Riddargatan 1.The design is a two-armed randomized controlled non-inferiority study, and outcomes are measured in terms of changes in alcohol consumption, problematic alcohol use, alcohol dependence alcohol use disorder, anxiety, as well as depression and quality of life. 600 participants are recruited online from the clinic's website. Consenting participants will complete baseline questionnaires online and participate in face-to-face assessment by a physician at the clinic. Eligible individuals will then be randomized into one of two groups: 1.Internet-based treatment program with online counselor support. 2. Face-to-face treatment with 5 individual counselor sessions at the clinic. Follow-up will be conducted online after 3, 6, 12 and 24 months in both groups.

ELIGIBILITY:
Inclusion Criteria:

* AUDIT-score ≥16 points and/or fulfilling at least 3 criteria of alcohol dependence (ICD-10)

Exclusion Criteria:

* Risk of severe withdrawal symptoms.
* Risk of suicide.
* Other psychiatric diagnosis that requires current treatment.
* Need for medication for alcohol dependence.
* Inadequate Swedish language skills.
* No Internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Time Line Follow Back (TLFB) | 3, 6, 12 and 24 months
  Change in number of standard drinks per day during last 7 days

SECONDARY OUTCOMES:
Time Line Follow Back (TLFB) Change in number of consumption days | 3, 6, 12 and 24 months
  Change in number of drinking days during last 7 days
Time Line Follow Back (TLFB) Change in number of days binge-drinking days | 3, 6, 12 and 24 months
  Change in number of binge-drinking days during last 7 days
Alcohol Use Disorders Identification Test Consumption (AUDIT-C) | 3, 6, 12 and 24 months
  Change in Quantity, Frequency and Binge-drinking scores during the time since last reported
Alcohol Use Disorders Identification Test (AUDIT) | 3, 6, 12 and 24 months
  Change in total AUDIT score, as a summarized measure of alcohol use since last reported
Montgomery Asberg Depression Rating Scale - Self report (MADRS-S) | 3, 6, 12 and 24 months
  Change in total MADRS-S score, as a summarized measure of depression
Generalised Anxiety Disorder Assessment (GAD-7) | 3, 6, 12 and 24 months
  Change in total GAD-7 score, as a summarized measure of anxiety
Questions about help-seeking behavior from family and friends | 3, 6, 12 and 24 months
  Change in help-seeking for alcohol related problems from family and friends. The questions about "other forms of support and treatment for problematic alcohol use during the trial period" were developed by our research group and used in a previous study of ours: Berman, A. H., Wennberg, P., & Sinadinovic, K. (2015). Changes in Mental and Physical Well-Being Among Problematic Alcohol and Drug Users in 12-Month Internet-Based Intervention Trials. Psychology of Addictive Behaviors, 29(1), 97-105. doi:10.1037/a0038420.PMID:25664387
Questions about help-seeking behavior from professionals | 3, 6, 12 and 24 months
  Change in help-seeking for alcohol related problems from professionals. The questions about "other forms of support and treatment for problematic alcohol use during the trial period" were developed by our research group and used in a previous study of ours: Berman, A. H., Wennberg, P., & Sinadinovic, K. (2015). Changes in Mental and Physical Well-Being Among Problematic Alcohol and Drug Users in 12-Month Internet-Based Intervention Trials. Psychology of Addictive Behaviors, 29(1), 97-105. doi:10.1037/a0038420.PMID:25664387

OTHER OUTCOMES:
The Readiness Ruler | 3, 6, 12 and 24 month
  Scores between 0 and 100. In this study, "How ready to change reduce my drinking" and "How ready to quit drinking".
Use of Internet-based program and website | From baseline to 3 months
  Number of visits and number of completed exercises in the Internet-based program and website
Session rating scale (SRS) | 2 and 5 weeks in to treatment
  4 scale questions on the user's alliance with the counselor
Working Alliance Inventory-Short Revised (WAI-SR) | 2 and 5 weeks in to treatment
  12 questions on working alliance adapted for Internet-based programs

CONTACTS AND LOCATIONS:
Overall Officials: Sven Andreasson, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Department of Public Health Sciences, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sinadinovic K, Wennberg P, Johansson M, Berman AH. Targeting individuals with problematic alcohol use via Web-based cognitive-behavioral self-help modules, personalized screening feedback or assessment only: a randomized controlled trial. Eur Addict Res. 2014;20(6):305-18. doi: 10.1159/000362406. Epub 2014 Oct 4. PMID 25300885
- See also: Clinic website — http://riddargatan1.se